CLINICAL TRIAL: NCT02150980
Title: INORMUS 40,000: Large Observational Cohort Study of Orthopedic Trauma Patients
Brief Title: INternational ORthopaedic MUlticenter Study in Fracture Care (INORMUS)
Acronym: INORMUS
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McMaster Surgical Associates (Other); National Health and Medical Research Council, Australia (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Mohit Bhandari, Professor of Surgery, Chair of Division of Orthopaedics, McMaster University
Other Study IDs: INORMUS_INTERNATIONAL
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Fractures or Dislocations
Keywords: Fractures; burden of fractures; orthopaedic fractures; orthopaedic injuries; orthopaedic trauma; observational study; outcomes of fracture care; epidemiology
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: Worldwide, injuries from trauma represent a major public health problem. The World Health Organization (WHO) has deemed this problem as one of the most important global priorities, calling 2011-2020 the 'Decade of Action for Road Safety'. Despite this, there is little empirical data in low and middle-income countries quantifying the burden of musculoskeletal injuries.

Methods: INORMUS is a global, prospective, multi-center, observational cohort study. The primary objective of the study is to determine the mortality, re-operation and infection rates of musculoskeletal trauma patients within 30 days post-hospital admission. The INORMUS study seeks to enroll 40,000 patients from low-middle income countries in Africa, Asia, and Latin America.

DETAILED DESCRIPTION:
Number of Participants:

40,000

Primary Research Objectives:

To determine among adult individuals admitted to hospital with musculoskeletal trauma (e.g. fractures or dislocations):

1. The incidence of major complications (mortality, re-operation and infection) as a composite outcome and the components of the composite within 30 days post-hospital admission.
2. The factors (system and patient variables) associated with the composite of major complications (mortality, re-operation and infection) within 30 days post-hospital admission.

Secondary Research Objective:

To determine the rates of major complications within 30 days post-hospital admission by type of fracture treatment provided (e.g. splinting versus operative fixation) and admission to hospital time (e.g. <72 hours or > 72 hours).

Diagnosis and Main Inclusion Criteria:

This study has minimal exclusion criteria by design. All patients 18 years of age or older admitted to a recruiting hospital for treatment of an orthopaedic injury that occurred within 3 months will be eligible for participation. Patients who are diagnosed with an orthopaedic fracture, dislocation, or fracture dislocation of the appendicular skeleton or spine will be included.

Study Outcomes:

The primary outcome is a composite of mortality, mortality, re-operation and infection within 30 days from hospital admission for all research objectives.

Duration of Patient Follow-Up:

Study participants will be followed until 30 days post hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older
* admitted to a recruiting hospital for treatment of an orthopaedic injury
* injury occurred within 3 months of hospital admission
* patients diagnosed with an orthopaedic fracture, dislocation, or fracture dislocation of the appendicular skeleton or spine will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 18 years of age or older who are admitted to a recruiting hospital in low-middle income countries in Africa, Asia, and Latin America
Sampling Method: Non-Probability Sample
Enrollment: 39797 (Actual)
Dates: Start 2014-04; Primary Completion 2023-11 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
mortality, re-operation and infection | 30 days post-hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, PhD, Principal Investigator — McMaster University; Philip Devereaux, MD, PhD, Principal Investigator — McMaster University; Rebecca Ivers, MPH, PhD, Principal Investigator — The George Institute
Locations (69):
- Clínica Zabala, Buenos Aires, Argentina
- Princess Marina Hospital, Gaborone, Botswana
- Brazil (2):
  - Hospital de Clínicas - UNICAMP, São José dos Campos
  - Hospital de Beneficencia Sirio-Libanes, São Paulo
- Baptist Hospital Mutengene, Mutengene, Cameroon
- China (14):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Anzhen Hospital affiliated to Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Beijing, Beijing Municipality
  - Xiamen University affiliated First Hospital, Xiamen, Fujian
  - Langfang Aidebao General Hospital, Langfang, Hebei
  - Langfang People's Hospital, Langfang, Hebei
  - Harbin Medical University Second hospital, Harbin, Heilongjiang
  - Second Bethune Hospital of Jilin University, Changchun, Jilin
  - Shenyang Orthopaedic Hospital, Shenyang, Liaoning
  - Hanzhong People's Hospital, Hanzhong, Shaanxi
  - Shanghai No.10 People's Hospital, Shanghai, Shanghai Municipality
  - Tianjin Hospital, Tianjin, Tianjin Municipality
  - The 2nd affiliated hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Colombia (2):
  - Centro Médico Imbanaco, Cali
  - Clinica Fracturas y Fracturas, Pereira
- Black Lion Hospital, Addis Ababa, Ethiopia
- Komfo Anokye Teaching Hospital (KATH), Kumasi, Ghana
- India (14):
  - Smt N H L Municipal Medical College, Gujrāt, Ahmedabad
  - Baptist Christian Hospital, Tezpur, Assam
  - St John Medical College, Bangalore
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - AIIMs Hospital, Delhi
  - Indian Institue for Spinal Care, Delhi
  - CMC Ludhiana, Ludhiana
  - Dr L H Hiranandani Hospital, Mumbai
  - Indira Ganghi Medical College, Puducherry
  - Medical College & Hospital, Bharati Vidyapeeth Deemed University, Pune
  - Noble Hospital, Pune
  - Sancheti Institute for Orthopaedics and Rehabilitation, Pune
  - CMC Vellore, Vellore
  - Data Meghe Institute of Medical Sciences, Wardha
- Sina Trauma and Surgery Research Center/University of Tehran, Tehran, Iran
- Kenya (4):
  - Rift Valley provincial hospital, Karuru One
  - Kiambu District Hospital, Kiambu
  - AIC Kijabe Hospital, Kijabe
  - Kenyatta National Hospital, Nairobi
- University of Malawi, Blantyre, Malawi
- Mexico (6):
  - Hospital Civil de Guadalajara, Guadalajara
  - Social Security Hospitals, Guadalajara
  - Hospital Puerta de Hierro, Jalisco
  - Social Security Hospitals, Mexico City
  - Social Security Hospital, Monterrey
  - Christus Muguerza Hospital Saltillo, Saltillo
- Lumbini Medical College, Kathmandu, Nepal
- Nigeria (2):
  - National Orthopaedic Hospital Enugu, Enugu
  - State trauma and surgical centre, Ondo
- Northwest General Hospital & Research Centre, Peshawar, Pakistan
- Hospital Santo Tomás, Panama City, Panama
- Instituto de Prevision Social - Central Hospital, Asunción, Paraguay
- Philippine General Hospital, Manila, Philippines
- University Teaching Hospital, Kigali, Rwanda
- South Africa (3):
  - Charlotte Maxete Johannesburg Acadamic Hospital, Johannesburg
  - Chris Hani Baragwanath Acadamic Hospital, Johannesburg
  - Helen Joseph Hospital, Johannesburg
- Tanzania (2):
  - Muhimbili Orthopaedic Institute, Dar es Salaam
  - Kilimanjaro Christian Medical Centre, Moshi
- Thailand (2):
  - Ramathibodi Hospital, Bangkok
  - Khon Kaen Hospital, Khon Kaen
- Uganda (2):
  - Fort Portal Regional Referral Hospital, Fort Portal
  - Mulago Hospital, Makerere University College of Health Sciences, Kampala
- Hospital Universitario de Caracas, Caracas, Venezuela
- Vietnam (2):
  - Viet Duc Hospital, Hanoi
  - Cho Ray Hospital, Ho Chi Minh City

REFERENCES:
- [Background] Mock C, Cherian MN. The global burden of musculoskeletal injuries: challenges and solutions. Clin Orthop Relat Res. 2008 Oct;466(10):2306-16. doi: 10.1007/s11999-008-0416-z. Epub 2008 Aug 5. PMID 18679760
- [Background] Fitzharris M, Zhong W, Myburgh J, Xuezhong Y, Yu J, Hammond N, Finfer SR, Taylor C, Wu Y. The status of trauma registry systems in Chinese hospitals. Inj Prev. 2011 Dec;17(6):419-21. doi: 10.1136/injuryprev-2011-040216. Epub 2011 Oct 13. PMID 21998256
- [Background] Fitzharris M, Yu J, Hammond N, Taylor C, Wu Y, Finfer S, Myburgh J. Injury in China: a systematic review of injury surveillance studies conducted in Chinese hospital emergency departments. BMC Emerg Med. 2011 Oct 26;11:18. doi: 10.1186/1471-227X-11-18. PMID 22029774
- [Background] Bhalla K, Harrison JE, Shahraz S, Fingerhut LA; Global Burden of Disease Injury Expert Group. Availability and quality of cause-of-death data for estimating the global burden of injuries. Bull World Health Organ. 2010 Nov 1;88(11):831-838C. doi: 10.2471/BLT.09.068809. Epub 2010 Jun 22. PMID 21076564
- [Background] Foote CJ, Petrisor B, Beyene J, Devereaux PJ, Dhillon M, Sancheti P Kotwal P, Miclau T, Bhandari M, and the INORMUS Investigators. International Orthopaedic Multicenter Fracture Study (INORMUS). Paper presented at: Orthopaedic Trauma Association 2012 Annual Meeting; 2012 October 3-6; Minneapolis, Minnesota.
- [Background] INORMUS Investigators. INternational ORthopaedic MUlticentre Study (INORMUS) in Fracture Care: Protocol for a Large Prospective Observational Study. J Orthop Trauma. 2015 Oct;29 Suppl 10:S2-6. doi: 10.1097/BOT.0000000000000404. PMID 26356208
- [Background] Foote CJ, Mundi R, Sancheti P, Gopalan H, Kotwal P, Shetty V, Dhillon M, Devereaux P, Thabane L, Aleem I, Ivers RQ, Bhandari M; INORMUS Investigators. Musculoskeletal trauma and all-cause mortality in India: a multicentre prospective cohort study. Lancet. 2015 Apr 27;385 Suppl 2:S30. doi: 10.1016/S0140-6736(15)60825-X. Epub 2015 Apr 26. PMID 26313078
- [Background] INORMUS Investigative Committee on behalf of all INORMUS Investigators. Operationalizing an orthopaedic research plan in the Decade of Action for Road Safety: the INternational ORthopaedic MUlticenter Study in Fracture Care. J Orthop Trauma. 2014;28 Suppl 1:S29. doi: 10.1097/BOT.0000000000000119. No abstract available. PMID 24857994
- [Derived] Pouramin P, Li CS, Busse JW, Sprague S, Devereaux PJ, Jagnoor J, Ivers R, Bhandari M; INORMUS investigators. Delays in hospital admissions in patients with fractures across 18 low-income and middle-income countries (INORMUS): a prospective observational study. Lancet Glob Health. 2020 May;8(5):e711-e720. doi: 10.1016/S2214-109X(20)30067-X. PMID 32353318
- See also: United Nations Global Road Traffic Safety Collaboration — http://www.who.int/roadsafety/en/
- See also: Canadian Orthopaedic Association: Call for Action Group — http://www.coa-aco.org/
- See also: WHO's Make Roads Safe Campaign — http://www.makeroadssafe.org/Pages/home.aspx
- See also: McMaster University International Surgery Desk — http://www.makeroadssafe.org/Pages/home.aspx